CLINICAL TRIAL: NCT00713882
Title: Health and Psychosocial Outcomes in Long-Term Lymphoma Survivors
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Carrie A. Thompson, M.D., Weill Cornell Medical College
Other Study IDs: 0802009649
Record Dates: First submitted 2008-07-07; First posted 2008-07-14 (Estimated); Last update posted 2009-03-12 (Estimated); Status verified 2009-03

CONDITIONS: Lymphoma, Non-Hodgkins; Hodgkins Disease
Keywords: Survivors; Quality of Life
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Hodgkin Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observational

SUMMARY:
The aims and objectives of this research are to identify chronic health conditions, psychological disease, quality of life issues, and patient preferences for survivorship care in patients who have survived aggressive lymphoma.

Subjects will be asked to participate in an oral interview with the primary investigator, either in-person or over the telephone. It is estimated that the survey will take about an hour.

DETAILED DESCRIPTION:
Survival rates for both non-Hodgkin's (NHL) and Hodgkin's lymphoma (HL) have improved in recent years due to the development of better treatments. However, the diagnosis and treatment may leave a cancer survivor with long-term consequences. It is recognized that patients cured of HL have increased mortality due to long-term effects of treatment. The literature also suggests that patients cured of NHL suffer from long-term complications. These complications may include infertility, cardiovascular disease, pulmonary disease, secondary cancer, osteoporosis, fatigue, and psychological disease. Limitations of the current literature on lymphoma survivors include that the majority of studies are retrospective in nature, and therefore do not take into account other risk factors for development of chronic health conditions, such as tobacco use, exercise, family history, and specifics of the cancer treatment. In addition, few studies have attempted to explore the relationship between chronic health conditions, psychological distress, patient-physician communication, and quality of life (QOL) in lymphoma survivors.

The aims and objectives of this research are to identify chronic health conditions, psychological disease, QOL, and patient preferences for survivorship care. A prediction model will then be developed integrating demographic, clinical, and health behavior data with chronic health conditions to predict poor psychosocial outcomes.

Subjects will be asked to participate in an oral interview with the primary investigator. The survey consists of demographic information, employment and workplace information, the Charlson Comorbidity Index, the Qualify of Life-Cancer Survivor questionnaire, the PHQ-9 (a depression screening tool), the Impact of Events Scale (a post-traumatic stress disorders screen), the State-Trait Anxiety Index, the Holmes-Rahe Stress Scale, Brief Fatigue Inventory, Leisure Time, Exercise Questionnaire, as well as questions pertaining to patient-physician communication and preferences for follow-up care. There are a series of qualitative or open-ended questions at the end of the survey, designed to understand the experience of being a survivor of lymphoma. These responses will be audio-taped (with the consent of the participant) in order to capture the verbatim responses of the participants, which is necessary for analysis of qualitative data.

Data will be entered into a password-protected database maintained by the primary investigator. Quantitative analysis will be done in JMP®7 statistical software. Analysis will be via multiple regression, with quality of life as the primary outcome. Predictive variables will include demographics, treatment data, comorbidities, fatigue, exercise, workplace issues, depression, anxiety, and post-traumatic stress disorder. Each variable will also be analyzed in a univariate model. Qualitative questions will be analyzed separately using grounded theory, a form of analysis that can be used to generate new ideas. This will involve selective coding technique, grouping concepts into categories, which lead to themes between the categories.

There are few risks involved with this study. It is possible that subjects may experience psychological distress due to the sensitive nature of some of the questions. In this case, participants may stop the interview at any time and withdraw consent. However, it is anticipated that this is unlikely to occur. In the event that the investigator finds that a subject has screened positive for depression, post-traumatic stress disorder, or anxiety; the patient's primary care physician will be notified, as long as the patient gives consent. If the patient is found to be suicidal at the time of the interview, the interviewer will accompany the patient to the emergency room.

Benefits of this research are the improved understanding of long-term outcomes in lymphoma survivors and the identification of factors that predict for poor QOL, so that in the future, interventions can be made to improve QOL in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* adults who have been treated for either aggressive lymphoma (Hodgkins lymphoma, diffuse large B-cell lymphoma, follicular grade III NHL, or others)
* are greater than 2 years from the time of last treatment
* no known active cancer

Exclusion Criteria:

* unable to participate in an interview in English
* indolent lymphoma (i.e. non-curable, including follicular grades 1-2 NHL)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be identified via physician referral at Weill Cornell Medical College, Hematology-Oncology outpatient clinic, or self-referral.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2008-04; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Quality of life | cross-sectional (time of interview)

CONTACTS AND LOCATIONS:
Overall Officials: Carrie A Thompson, M.D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States